CLINICAL TRIAL: NCT06912828
Title: Whole Genome Association Study (GWAS) to Identify Predictive Genetic Factors for the Success of Dietary Intervention in the Treatment of Irritable Bowel Syndrome (IBS) Symptoms
Brief Title: GWAS to Identify Predictive Genetic Factors for the Success of Dietary Intervention in the Treatment of IBS Symptoms
Status: Recruiting | Type: Observational
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Arezina Kasti, PhD candidate - Head of Clinical Nutrition Department of Attikon Hospital, Attikon Hospital
Other Study IDs: ΕΒΔ407/30.5.2024
Record Dates: First submitted 2025-01-14; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Irritable Bowel Syndrome (IBS); Genome-wide Association Study; Single Nucleotide Polymorphisms; Mediterranean Diet; FODMAP Diet
Keywords: diet response; nutrigenetics
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Basic group: MED-LFD Diet for 2 - 6 weeks. After this period there will be a reintroduction phase protocol that will last 6 - 8 weeks.
  Interventions: Other: Med-LFD intervention

INTERVENTIONS:
Other: Med-LFD intervention — In the beginning of the intervention, blood and stool samples will be collected. All participants of the group at phase 1 (elimination phase), will initially follow the Med- LFD (2-6 weeks). At phase 2 (reintroduction phase), patients will gradually reintroduce foods rich in FODMAPs (6-8 weeks) and test their tolerance. At phase 3 (maintenance phase), following the reintroduction of foods rich in FODMAPs, patients will follow an individualized diet based on their personal tolerance (a combination of high and low FODMAPs). In the end of intervention, stool samples will be collected again.

SUMMARY:
This is a GWAS that aims to identify possible single nucleotide polymorphisms (SNPs) that are associated with the response in a combined dietary pattern low in fermentable oligosaccharides, disaccharides, monosaccharides, and polyols and Meditteranean diet (MED-LFD) in a small group of patients with Irritable Bowel Syndrome (IBS).

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a very common chronic gastrointestinal disorder. Several factors seem to contribute to its development, such as psychological stress, intestinal dysbiosis, infections, post-traumatic syndrome and genetic predisposition. Regarding the nutritional management of IBS, there are several approaches to alleviate symptoms, such as the low-fructose diet low in fermentable oligosaccharides, disaccharides, monosaccharides and FODMAP polyols (LFD), recommendations from the British Institute of Health and Care Excellence (NICE) and the recently proposed combination of the Mediterranean diet and LFD (MED-LFD) proposed by our Research Group. However, genetic background expressed in single nucleotide polymorphisms (SNPs) appears to influence the response to even dietary interventions.

The aim of this GWAS is to identify SNPs that are associated with the negative or positive response to the diet.

At the baseline, blood samples will be collected for DNA extraction. Genotyping will be based on Next Generation Sequencing (NGS) technology to detect genetic factors associated with the effectiveness of the intervention. Symptom severity will be measured by the IBS-SSS scale. Mental health status will be assessed with the HADS (Hospital Anxiety and Depression Scale) questionnaire.

Patients will be recruited by the Department of Clinical Nutrition, Attikon University General Hospital, where the nutritional intervention will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of the Rome IV criteria for IBS
* Provision of written informed consent.
* Commitment of availability throughout the study period.
* IBS-SSS > 175

Exclusion Criteria:

* Any concomitant disease requiring specialized nutrition (e.g. renal failure, diabetes, celiac disease, cerebrovascular disease of the central nervous system, major surgical cavity).
* Pregnancy.
* Breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18-65 years with IBS (fullfiling ROME IV criteria) who have IBS-SSS>175. People with any concomitant disease requiring specialized nutrition, pregnant or lactating women will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Find single nucleotide polymorphisms (SNPs) that associate with the diet respone | Baseline
  Blood samples will be collected for DNA extraction. Genotyping be based on Next Generation Sequencing (NGS). Quality control (QC) filtering will be applied at individual-and variant-level using specialized software.

SECONDARY OUTCOMES:
Change of symptoms severity pre and post intervention using a specialized questionnaire. | Baseline and through study completion (an average of 1 year)
  IBS- SSS contains 5 specific questions with instructions on how to score them. Each of the five questions (pain severity, pain frequency, abdominal distension severity, bowel movement satisfaction, quality of life) ranges from 0 to a maximum score of 100 using a visual analog scale (VAS) with total scores ranging from 0 to 500, with higher scores indicating more severe symptoms. Subjects can be categorized as having mild (75-175), moderate (175-300), or severe (>300) IBS. A decrease of 50 points is associated with a clinically meaningful improvement.
Evaluation of the effect of interventions on gut microbiota composition between groups. | Baseline and through study completion (an average of 1 year)
  Fecal samples will be collected from each participant and stored at -80°C.
Assessment of general quality of life pre and post intervention between groups | Baseline and through study completion (an average of 1 year)
  12-Item Short Form Survey (SF-12) is a 12-item questionnaire used to assess generic health outcomes from the patient's perspective, covering the eight domains of health outcomes: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional & mental health. The items are weighted and summed to provide physical and mental health scores (PCS and MCS). The two composite scores are computed using the scores on the questions that range from 0 to 100, with higher score indicating better health.
Assessment of symptoms burden in general pre and post intervention. | Baseline and through study completion (an average of 1 year)
  The GSRS questionnaire was originally developed for dyspeptic patients but was later validated in patients with IBS. The GSRS is a 15-item questionnaire designed to assess common gastrointestinal symptoms. The questionnaire has five subscales, reflux, diarrhea, constipation, indigestion, and abdominal pain, with subscale scores ranging from 1 (no discomfort) to 7 (severe discomfort). Higher scores represent higher symptom burden.
Assessment of anxiety and depression disorders pre and post intervention. | Baseline and through study completion (an average of 1 year)
  The Hospital Anxiety and Depression Scale (HADS) questionnaire is used for the assessment of anxiety and depression symptoms. It's a 14-item scale with seven items for each subscale, anxiety (HADS-A) and depression (HADS-D). Each item is scored on a response scale with four alternatives, ranging between 0 and 3. The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). A final score of 0-7 on each scale indicates that the patient has no symptoms, a score of 8-10 indicates mild symptoms while a score ≥11 indicates severe symptoms of anxiety and depressive disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Attikon General University Hospital of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: No